CLINICAL TRIAL: NCT06410053
Title: The All Ireland Infectious Diseases Cohort Project - AIID Cohort Project
Brief Title: The All Ireland Infectious Diseases Cohort Project
Acronym: AIID
Status: Recruiting | Type: Observational
Sponsor: University College Dublin (Other)
Collaborators: Beaumont Hospital (Other); Children's Health Ireland (Other Government); Cork University Hospital (Other); Mater Misericordiae University Hospital (Other); Our Lady of Lourdes Hospital, Drogheda (Other Government); St. James's Hospital, Ireland (Other); St. Luke's Hospital, Ireland (Other); St Vincent's University Hospital, Ireland (Other); Wexford General Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: AIID Cohort
Record Dates: First submitted 2023-04-05; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Infectious Disease
Keywords: Human Immunodeficiency virus; COVID-19; Viral hepatitis; Skin and soft tissue infections; Bone infection
MeSH Terms: conditions — Communicable Diseases; Acquired Immunodeficiency Syndrome; COVID-19; Soft Tissue Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood sample to be prepared as plasma, serum and viable peripheral blood mononuclear cells (PBMC) for cryopreservation.
  2. Respiratory samples (where relevant e.g., subject with respiratory viral infection or pulmonary TB)
  3. Stool sample for later microbiome analysis (optional)
  4. Urine
  5. Swabs, including mucosal (e.g., ano-genital, naso-pharyngeal) and superficial (skin).
  In addition, where subjects undergo lumbar puncture testing as part of routine care, any excess available sample may also be stored.
  These stored samples provide the opportunity for future research studies investigating host factors associated with the response to infection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The All-Ireland Infectious Diseases (AIID) Cohort is a multicentre, prospective, longitudinal observational cohort that enrols consecutive adult subjects attending participating institutions for infectious disease services. This is an ongoing prospective observational cohort of unlimited duration.

DETAILED DESCRIPTION:
The All-Ireland Infectious Diseases cohort study (AIID Cohort) is enrolling patients at a number of Irish Hospitals with infectious diseases, including Covid-19. The AIID Cohort is a multicentre, prospective, longitudinal, observational cohort that enrols consecutive adult subjects (>18 years old) attending hospitals services for management of infections.

Subjects provide consent for use of routine clinical and laboratory data for research. All data is collected by a combination of retrospective medical note review and extraction of data from electronic health records. At a minimum, the following data items are to be collected at enrolment and subsequent clinic visits:

1. Demography and basic information (e.g. date of birth, gender, country of origin, ethnicity, anthropometric assessments, and reasons for the attendance, date or year for disease diagnosis and transmission risk.
2. Laboratory data: Relevant routine virological (including genotyping) and immunological data for characterisation of the HIV infection, TB, hepatitis C, COVID-19 and other relevant co-infections will also be collected as well as other relevant clinical routine data on tolerability and safety (i.e., renal, liver, lipids)
3. Medical treatment: All medications, including start-and stop dates and reason for discontinuation, adherence. Concomitant medical treatment related to co-infections and co-morbidities.
4. Clinical events: hospitalisation, diseases specific relevant active and previous diagnosis (e.g., AIDS and non-AIDS events, including comorbidities).

In addition, subjects are asked to provide biological samples for up to five occasions every six months for bio-banking for host profiling and pathogen bio-repository. To provide flexibility for participants around requirements for fasting or scheduling, participants may be asked to attend to provide samples for biobanking outside of routine scheduled clinic visits. These stored samples provide the opportunity for future research studies investigating host factors associated with the response to infection.

The AIID Cohort is approved by local institutional review boards and all participants provide written, informed consent. Data and samples within the AIID Cohort are accessed through standardised Data Access Guidelines and all approved Data Access Requests are approved by the local Ethics Committee.

ELIGIBILITY:
Inclusion criteria:

* ≥ 18 years of age patients attending clinical services of participating institutions with issues related to infectious diseases.
* Willing and able to provide informed consent or
* Provide deferred assent if an incapacitated or unconscious patient is unable to provide informed consent

Exclusion criteria:

* Patients under 18 years of age
* Patients with learning disabilities, mental illness, or dementia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients attending Clinical Services relating to infectious diseases at participating hospitals in Ireland who provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Establishment of data rich cohort | through study completion, an average of 1 year
  Overall number of recruited participants and number of recruited participants with major conditions (COVID-19, HIV, TB)

SECONDARY OUTCOMES:
Cohort retention | through study completion, an average of 1 year
  Number of subjects in care or mortality
Cohort associated metadata | through study completion, an average of 1 year
  Number of subjects recruited to the cohort with completed metadata and biobanked samples

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Mallon, PhD, FRCPI, Principal Investigator — UCD
Locations (9):
- Ireland (9):
  - Cork University Hospital, Cork
  - Our Lady of Lourdes Hospital, Drogheda, Drogheda
  - St Vincent's University Hospital, Ireland, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Children's Health Ireland at Crumlin, Dublin
  - St James's Hospital, Dublin
  - St Luke's General Hospital, Kilkenny, Kilkenny
  - Wexford General Hospital, Wexford

REFERENCES:
- See also: AIID Cohort Project — https://www.ucd.ie/medicine/research/researchcentres/ucdcentreforexperimentalpathogenhostresearch/allirelandinfectiousdiseasescohortstudy/